CLINICAL TRIAL: NCT03857061
Title: COPDwear V2 - A Wearable and a Self-management Application for COPD Patients at Home: a Pilot Prospective Cohort Study
Brief Title: A Wearable and a Self-management Application for Chronic Obstructive Pulmonary Disease (COPD) Patients at Home
Acronym: COPDwear
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other); Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Robert Wu, General Internal Medicine Site Director, University Health Network, Toronto
Other Study IDs: 18-5462
Record Dates: First submitted 2018-07-23; First posted 2019-02-27 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: wearables; self-monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD Patients: This is a prospective cohort study enrolling patients with COPD to 1) wear a smartwatch that passively senses heart rate, motion, audio, 2) use a smartphone that can obtain oxygen saturation upon demand, 3) use a self-management app on the smartwatch, smartphone and a webapp.
  Interventions: Device: smartphone, smartwatch, WearCOPDv2 application

INTERVENTIONS:
Device: smartphone, smartwatch, WearCOPDv2 application — WearCOPD2 consists of hardware and software components.
  6.1 Hardware The hardware for wearCOPDv2 consists of three main components; (1) a smartwatch, (2) a phone, and (3) a server.
  6.2 Software
  The wearCOPDv2 system has two main software components:
  1. Data collection service
  2. Participant user interface

SUMMARY:
Our overall research goal for this project is to create a wearable device and mobile application, appealing to patients with Chronic Obstructive Pulmonary Disease (COPD), which provides them with appropriate self-management tools and detects AECOPDs early to permit prompt treatment and prevent severe exacerbations requiring hospitalization.

DETAILED DESCRIPTION:
Our overall research goal for this project is to create a wearable device and mobile application, appealing to patients with COPD, which provides them with appropriate self-management tools and detects Acute Exacerbations of COPD (AECOPDs) early to permit prompt treatment and prevent severe exacerbations requiring hospitalization. Currently, the investigators are developing a second version of this app, WearCOPDv2. This app will incorporate features identified as being desirable from our patient interviews: 1) new sensor that was requested by patients - oxygen saturation, and 2) the app will incorporate a patient-facing interface as patients requested a method to view their data as well as access to information to learn how to manage their condition better.

Research questions:

Can an app designed for patients with COPD that includes biosensor feedback improve self-management of COPD?

What is the accuracy of our sensor data (heart rate, activity, respiratory rate, oxygen saturation, coughing, and other sounds of interest) in detecting early AECOPDs?

ELIGIBILITY:
Inclusion Criteria:

* Able to speak English
* Moderate to very severe COPD (GOLD C and D) as defined by the GOLD guidelines
* Clinically relevant disease, as defined by a history of exacerbation in the previous 12 months
* Previous spirometry or Pulmonary Function Test results of Forced Expiration Volume/Forced Vital Capacity (FEV1/FVC) <0.70 with an FEV1 below 80% predicted
* Patient resides at home (not long term care residence or another hospital)

Exclusion Criteria:

* Pulmonary condition other than COPD as the main respiratory disease such as bronchiectasis or asthma
* Rapid lethal disease, e.g. lung cancer, advance heart failure, end-stage renal disease
* Any medical conditions that would impair their ability to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit patients who have clinically relevant COPD who live at home. They will be identified in clinics and the wards by members of their care team. Posters informing people of the study will also be posted at University Health Network (UHN) with a contact number.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in self-management as measured by the Mastery sub-section of the Chronic Respiratory Disease Questionnaire | 6 months
  Can an app designed for patients with COPD that includes biosensor feedback improve self-management of COPD?
  We will use the Mastery sub-section of the Chronic Respiratory Disease Questionnaire to measure our research question. Mastery is measured with a 7-point likert scale where higher scores indicate better health-related mastery.

SECONDARY OUTCOMES:
Change in self-efficacy as measured by the COPD Self-Efficacy Scale | 6 months
  Can an app designed for patients with COPD that includes biosensor feedback improve self-efficacy of COPD?
  This will be measured by the COPD self-efficacy scale. Participants will determine how confident they are that they could manage breathing difficulty or avoid breathing difficulty in certain situations. Usin the following scale.
  1. Very confident
  2. Pretty confident
  3. Somewhat confident
  4. Not very confident
  5. Not at all confident
  A lower score indicates higher self-efficacy.
Change in Health related quality of life as measured by the St. George's respiratory questionnaire | 6 months
  Can an app designed for patients with COPD that includes biosensor feedback improve health related quality of life?
  Scoring and Scales
  Questions 1 - 7 Scale: Most days a week - Not At All
  Where a patient has ticked a box, a value of 1 is entered for the appropriate question.
  Question 8 Where a patient has ticked 'Yes' to having a worse wheeze in the morning, a value of 1 is entered for the appropriate question.
  Questions 9, 10 & 17 Where a patient has ticked a box, a value of 1 is entered for the appropriate question.
  Questions 11 - 16 Where a patient has ticked 'True' a value of 1 is entered for the appropriate question.
  In response to question 14, if a patient is not receiving medication, enter the responses as zero.
  Score = 100 x (Summed weights from positive items in the questionnaire divided by the Sum of weights for all items in the questionnaire)
  lower scores indicate higher health related quality of life
Change in symptom scale as measured by the MRC dyspnea scale | 6 months
  Can an app designed for patients with COPD that includes biosensor feedback improve COPD symptoms?
  The MRC Dyspnea scale asks you to rate your breathlessness on a 5 point likert scale.
Accuracy of our derived prediction algorithm to detect acute exacerbations as measured by the daily symptom score. | 6 months
  We will correlate sensor data from the smartwatch to exacerbations defined by the daily symptom score.
  The daily symptom score asks about daily symptoms of COPD and patients are asked to answer yes or no to whether or not they have experienced a decline of any of the symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wu, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
UHN, research personnel will have direct access to the source documents with identifying information.
  UHN, University of Toronto (UofT) and Samsung Research America (SRA) will have access to the anonymized subject data for analysis purposes.
Supporting Information: Study Protocol
Time Frame: Data will become available right away for up to 5 years.
Access Criteria: Data will be stored and analyzed on the secure UHN server

REFERENCES:
- [Derived] Wu R, de Lara E, Liaqat D, Liaqat S, Chen JL, Son T, Gershon AS. Feasibility of a wearable self-management application for patients with COPD at home: a pilot study. BMC Med Inform Decis Mak. 2024 Mar 5;24(1):66. doi: 10.1186/s12911-024-02461-y. PMID 38443858